CLINICAL TRIAL: NCT04655261
Title: Prospective Multi-Center Observational Study to Assess Effectiveness of Venclexta (Venetoclax) in Combination With Obinutuzumab in Population of Previously Untreated Chronic Lymphocytic Leukemia Patients in Routine Clinical Practice in Russian Federation (FIRST)
Brief Title: Study of Oral Venetoclax Tablets in Combination With Intravenous Obinutuzumab Injection to Assess Achievement of Best Response in Adult Participants With Chronic Lymphocytic Leukemia
Acronym: FIRST
Status: Terminated | Type: Observational
Why Stopped: Lack of Recruitment
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-486
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Chronic Lymphocytic Leukemia (CLL); Venetoclax; Venclexta; Obinutuzumab; Cancer
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Treated With Venetoclax + Obinutuzumab: Participants will receive venetoclax (Venclexta) in combination with Obinutuzumab according to local label.

SUMMARY:
Chronic Lymphoid Leukemia (CLL) is the most common type of leukemia (cancer of blood cells) in adults affecting men more so than women. The main objective of this study is to assess the how effective venetoclax (Venclexta) in combination with Obinutuzumab is in treating Chronic Lymphocytic Leukemia (CLL). Effectiveness is assessed by achievement of best response.

Venetoclax is an approved drug developed for the treatment of CLL. Approximately 50 adult participants with previously untreated CLL will be enrolled in approximately 10 to 15 sites in Russian Federation.

Participants will receive oral venetoclax tablets in combination with intravenous (IV) Obinutuzumab as prescribed by the physician prior to enrolling in this study in accordance to the local practice and label.

There may be a higher burden for participants in this study compared to standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of previously untreated Chronic Lymphocytic Leukemia (CLL).
* Participant for whom the physician has decided to initiate CLL treatment with Venetoclax combo therapy with Obinutuzumab, according to approved local label up to 4 weeks (28 days) after Obinutuzumab treatment initiation.

Exclusion Criteria:

* Contraindications to Venclexta (Venetoclax) as listed on the approved local label in Russian Federation.
* Creatinine Clearance < 30 milliLitres/minute.
* Richter syndrome or Transformation of CLL to aggressive non-Hodgkin lymphoma.
* Participating in a clinical trial with an investigative drug for CLL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with previously untreated chronic lymphocytic leukemia (CLL)
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Overall Response Rate (ORR) Best Response | Up to approximately 36 Months
  ORR is defined as complete remission (CR) + complete remission with incomplete bone marrow recovery (CRi) + partial remission (PR) + nodular partial remission (nPR).

SECONDARY OUTCOMES:
Percentage of Participants Achieving Objective Response Rate (ORR) | Up to 12 Months
  ORR is defined as CR + CRi + PR + nPR.
Time to First Response | Up to approximately 36 Months
  Time to first response is defined as number of days from first venetoclax intake to first response.
Time to Best Response | Up to approximately 36 Months
  Time to best response is defined as number of days from first venetoclax intake to best response (CR, CRi, PR, nPR).
Duration of Response (DoR) | Up to approximately 36 Months
  Duration of Response (DoR) is defined as number of days from first response to disease progression or death from any cause, whichever comes first.
Time to Next Treatment | Up to approximately 36 Months
  Time to next treatment is defined as number of days from first venetoclax intake to first intake of next treatment including death from any cause.
Minimal Residual Disease (MRD) | Up to 36 Months
  Percentage of participants achieving MRD (CLL < 10000 leucocytes) in the bone marrow, peripheral blood, either and both will be assessed.
Overall Survival (OS) | Up to 36 Months
  OS is defined as the number of days from the date of first dose to the date of the observational period end or death for all dosed participants.
Progression-Free Survival (PFS) | Up to 36 Months
  PFS is defined as the interval (in days) between the first treatment day to the first sign of disease progression or death from any cause.
Number of Participants With Adverse Events (AEs) | Up to approximately 36 Months
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- Russia (4):
  - Moscow State budget healthcare /ID# 226058, Moscow, Moscow
  - Regional Children's Clinical Hospital of Volgograd /ID# 238328, Volgograd, Volgograd Oblast
  - Russian Research Institute of Hematology and Transfusiology of the FMBA /ID# 231127, Saint Petersburg
  - Tula Regional Clinical Hospital /ID# 231128, Tula

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-486&Latitude=&Longitude=&LocationName=#additional-resources-section